CLINICAL TRIAL: NCT05739201
Title: Comparative Study Between Interscalene Nerve Block, Anterior Suprascapular Nerve Block, and Pericapsular Nerve Group Block for Arthroscopic Shoulder Surgery
Brief Title: ISB, SSNB, and PENG Block for Arthroscopic Shoulder Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Shrouk Elsawaf, Resident, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 36264MS18/1/23
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Interscalene Nerve Block; Anterior Suprascapular Nerve Block; Arthroscopic Shoulder Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (I) (Active Comparator): 30 patients will receive interscalene nerve block.
  Interventions: Procedure: interscalene nerve block
- Group (II) (Active Comparator): 30 Patients will receive anterior suprascapular nerve block.
  Interventions: Procedure: anterior suprascapular nerve block
- Group (III) (Active Comparator): 30 atients will receive pericapsular nerve group block around shoulder surgery
  Interventions: Procedure: Peri-capsular nerve group block

INTERVENTIONS:
Procedure: interscalene nerve block — Patients will receive interscalene nerve block, in which the patient will be in supine position with the head turned to the contralateral side using an ultrasound scan to identify the C5 and C6 nerve roots between the scalene muscles.15 ml of 0.25% Bupivacaine will be deposited between the C5 and C6 nerve roots, within the interscalene groove using a 22 gauge-regional block needle.
  Arms: Group (I)
Procedure: anterior suprascapular nerve block — Patients will receive anterior suprascapular nerve block, in which the patient will be in supine position with the head turned to the contralateral side, using an ultrasound the nerve will be traced as it diverges from the brachial plexus to lie under the omohyoid muscle in the supraclavicular fossa. 15 ml of 0.25% Bupivacaine will be deposited lateral to the suprascapular nerve, underneath the omohyoid muscle using a 22 gauge-regional block needle.
  Arms: Group (II)
Procedure: Peri-capsular nerve group block — Patients will receive PENG block, in which the patient will be in supine position and the patient's arm will be placed in external rotation and abducted at 45 degrees, using an ultrasound the humeral head, the tendon of the subscapularis muscle and the deltoid muscle over it will be defined, 15 ml of 0.25% Bupivacaine will be placed between the deltoid muscle and subscapularis tendon using a 22 gauge-regional block needle.
  Arms: Group (III)

SUMMARY:
This study is designed to investigate the post-operative analgesic effect of interscalene nerve block or anterior suprascapular nerve block compared to pericapsular nerve group block in patient undergoing elective arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
Shoulder arthroscopy is a common outpatient operation with an increasing number of indications and complexity. Early postoperative pain immediately following shoulder surgery is a major concern and cause of distress for patients and orthopedic surgeons. Adequate pain control is vital for all aspects of the patient's recovery.

Nowadays, several ultrasound -guided regional anesthesia methods are used for postoperative analgesia. Regional techniques such as interscalene and supraclavicular blocks are usually preferred for shoulder analgesia. Interscalene brachial plexus block (ISB) is the gold standard technique in this area.

Suprascapular nerve block (SSB) has been proposed as an alternative to the ISB in providing analgesia for shoulder surgeries as it has a lower likelihood of causing phrenic nerve blockade.

The pericapsular nerve group (PENG) block has been suggested to be safely applied for analgesia and can be part of surgical anesthesia, but alone is not sufficient for anesthesia in shoulder surgery. The block of this area did not cause motor block or pulmonary complications, nor result in muscle laxity, blocking only the shoulder and the upper third of the humerus.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients.
* ASA class I and II and scheduled for elective shoulder arthroscopy.

Exclusion Criteria:

* Patient who refuses the regional anesthesia technique.
* History of allergy to local anesthetics.
* Local infection at the site of the block.
* History of Pre-existing major organ dysfunction such as hepatic and renal failure.
* History of pre-existing lung disease (COPD, uncontrolled asthma).
* Preexisting upper extremity neurological abnormality or neuropathy.
* Difficulties in comprehending (NRS).
* Chronic opioid users (opioid intake more than 3 months).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
the total opioid consumption. | 24-hour postoperatively
  Postoperative analgesia will be assessed by total opioid consumption and time till administration of first rescue analgesia will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ayman A Youssef, MD, Principal Investigator — Professor of Anaesthesiology, Surgical Intensive Care and Pain Therapy, Faculty of Medicine, Tanta University, Egypt
Locations (1):
- Shrouk Mohamed Elsawaf, Tanta, EL-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the principal investigator
Supporting Information: Study Protocol, SAP
Time Frame: one year